CLINICAL TRIAL: NCT05660057
Title: Evaluation of a New Computer Screen for Patients With Persisting Concussion Symptoms Including Computer Screen Intolerance.
Brief Title: Testing of a New Computer Screen for Patients With Persistent Concussion Symptoms (PCS).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 22-5525
Record Dates: First submitted 2022-12-02; First posted 2022-12-21 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Post-Concussion Symptoms
MeSH Terms: conditions — Post-Concussion Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will read a short story and watch moving images for 30 minutes or until any of their persisting concussion symptoms will arise on the standard computer monitor and the newly designed computer monitor in two visits.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Newly designed computer monitor (Experimental): Participants will read a short story and then watch moving images for 30 minutes or until any of their persisting concussion symptoms arise. The number and severity of symptoms will be assessed by completing SCAT -III pre- and post-study tasks.
  Interventions: Device: New computer monitor
- Standard computer monitor (Sham Comparator): Same participants will read a short story and watch moving images for 30 minutes or until any of their persisting concussion symptoms arise on the standard computer screen.The number and severity of symptoms will be assessed by completing SCAT -III pre- and post-study tasks.
  Interventions: Device: New computer monitor

INTERVENTIONS:
Device: New computer monitor — The device to be studied is a newly designed computer monitor and will be compared with the standard computer monitor.

SUMMARY:
This study will examine whether a newly designed monitor for computers is better tolerated by concussed patients than the standard computer monitor. The information gathered from this study will contribute to the understanding of the persisting concussion symptoms including computer screen intolerance and photosensitivity, with the aim of helping those with concussions.

DETAILED DESCRIPTION:
The study will involve completing a reading task on the standard computer monitor and the newly designed computer monitor. First, participants will be asked to rate their pre-test symptoms using a SCAT-III symptom checklist. Then they will read a short story and watch moving images on one of the devices (standard computer monitor or the newly designed computer monitor) for 30 minutes or until persisting concussion symptoms of moderate severity arise. Then, they will be asked to rate their post-test clinical symptoms using a SCAT-III symptom checklist. On a second visit, 7 to 10 days later, they will do the same activity on the other device. Each visit will take 60 minutes.

The study will involve 100 patients with a history of concussion and computer screen intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of persisting concussion symptoms (1 month to 5 year since concussion)
* Must speak English
* Must provide written consent
* No alcohol/recreational drug use within 24 hours of intervention
* No other neurological, psychiatric or ocular conditions

Exclusion Criteria:

* No diagnosis of Persisting Concussion Symptoms
* Under the age of 18, over the age of 65
* Other neurological/psychiatric or ocular conditions
* Alcohol or recreational drug use within 24 hours of intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
The investigators believe that patients will subjectively perceive the new monitor to be a more effective reading device than the standard monitor. | Two visits 7 to 10 days apart
  SCAT-III Symptoms checklist will be completed before and after study tasks (reading an excerpt and watching a moving image) to measure symptoms number and severity arising after the study task on a standard monitor and compare it to the newly designed monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Tator, MD, PhD, Principal Investigator — University Health Network, Toronto; Carmela Tartaglia, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Canadian Concussion Centre- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No